CLINICAL TRIAL: NCT07243509
Title: Evaluation of the Efficacy of Sliding Mechanisms on Round Versus Rectangular Archwires in Canine Retraction After First Premolar Extraction in Class II Malocclusion: A Randomized Clinical Trial
Brief Title: Evaluating the Efficacy of the Sliding Mechanisms on Round-section Arch Wire
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-2025-Ortho-10
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: CLASS II DIVISION 1 MALOCCLUSION
Keywords: Canine retraction; acceleration of orthodontic tooth movement; Bidimensioanl archwire; Sliding mechanics
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Canine retraction on a round cross-section archwire (Experimental): The patients in this group will be treated by sliding on a round cross-section archwire of 0.020-inch diameter.
  Interventions: Procedure: Round-cross-section archwire
- Traditional canine retraction on a rectangular-cross-section archwire (Active Comparator): The patients in this group will be treated using a sliding rectangular arch wire with a diameter of 0.019 × 0.025 inches.
  Interventions: Procedure: Rectangular-cross-section archwire

INTERVENTIONS:
Procedure: Round-cross-section archwire — Canines will be retracted on an archwire with a diameter of 0.20 inches.
  Arms: Canine retraction on a round cross-section archwire
Procedure: Rectangular-cross-section archwire — Canines will be retracted on an archwire with a diameter of 0.019 x 0.025-inch.
  Arms: Traditional canine retraction on a rectangular-cross-section archwire

SUMMARY:
Patients at the Orthodontic Department of the University of Damascus Dental School will be examined, and subjects who meet the inclusion criteria will be included. Then, initial diagnostic records (diagnostic gypsum models, internal and external oral photographs, and radiographic images) will be studied to ensure that the selection criteria are accurately matched.

This study aims to compare two groups of patients with mild to moderate skeletal Class II malocclusion (ANB angle between 5° and 7°), a normal to slightly increased vertical growth pattern (Björk's sum > 390° and < 406°), and an overjet of 5-10 mm. Experimental group: the patients in this group will be treated in the canine retraction phase with a sliding on a round-section archwire of 0.020 inch Control group: the patients in this group. Maxillary canine distalization was carried out using sliding mechanics on a 0.019 × 0.025-inch stainless steel archwire.

DETAILED DESCRIPTION:
In adult Class II camouflage treatment, the extraction of the first premolars is followed by a two-phase retraction protocol, consisting of initial canine retraction and subsequent incisor retraction, which is a standard approach. However, this process often extends treatment duration up to 36 months, creating significant clinical challenges. Prolonged orthodontic therapy not only burdens patients but also increases the risk of complications such as dental caries, root resorption, and periodontal problems, emphasizing the need for more efficient treatment strategies.

To accelerate tooth movement, both surgical and non-surgical methods have been explored. Surgical interventions, including corticotomy, piezocision, flapless cortico-alveolar perforations, and periodontal accelerated osteogenic orthodontics, have shown promising results but remain invasive and less acceptable to patients. Consequently, non-surgical alternatives have gained attention, including low-level laser therapy, electrical stimulation, platelet-rich plasma injections, and mechanical innovations such as self-ligating brackets. Despite these advances, canine retraction remains biomechanically demanding due to its slow rate and the difficulty of controlling unwanted rotation and angulation.

Mechanically, rectangular archwires provide torque control but generate high friction at the bracket-wire interface, delaying canine movement. Round-section archwires, by contrast, reduce bracket-wall contact and friction, enabling smoother sliding mechanics, improved angulation control, and reduced anchorage strain. Despite these theoretical advantages, clinical evidence is scarce. The only notable study, by Hamid, was limited by methodological shortcomings, including a short four-week observation period and a lack of long-term data. Importantly, no clinical trial has systematically evaluated sliding mechanics using a 0.020-inch round archwire, leaving a critical gap in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-25 years
* Mild to moderate skeletal Class II malocclusion (ANB angle between 5° and 7°),
* A normal to slightly increased vertical growth pattern (Björk's sum > 390° and < 406°),
* An overjet of 5-10 mm.
* A further prerequisite was a camouflage treatment plan involving the extraction of the maxillary first premolars.

Exclusion Criteria:

* the presence of no systemic health issues or any systemic condition known to influence the rate of orthodontic tooth movement,
* active periodontal disease,
* absence of any permanent teeth in the upper arch (excluding third molars),
* crowding of 4 mm or greater,
* inadequate oral hygiene.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Change in the Rate of Maxillary Canine Retraction | T0: 10 minutes before starting canine retraction stage; T1: 30 days following the onset of canine retraction; T2: 60 days; T3: 90 days following canine retraction onset; TF: At completion of canine retraction (expected to occur within 3-5 months)
  Canine displacement is measured by projecting the canine apex and the medial end of the third palatal ruga onto the mid-palatal plane; the linear distance between these points is recorded at each time point. Monthly retraction rates are calculated by dividing the change in displacement by the corresponding interval in months. For each subject, mean monthly rates for right and left canines are determined, and the cohort retraction rate is expressed as the average across all patients.

SECONDARY OUTCOMES:
Change in Canine Rotation | T0: 10 minutes before starting canine retraction stage; T1: 30 days following the onset of canine retraction; T2: 60 days; T3: 90 days following canine retraction onset; TF: At completion of canine retraction (expected to occur within 3-5 months)
  Canine rotation is defined as the angle between the mid-palatal plane and the line connecting the mesial and distal ridges of the canine crown. The angular shift between consecutive intervals is divided by the interval duration to yield monthly rotation rates. Per-subject averages for right and left canines are computed and then averaged across participants.
Change in Anchorage Loss | T0: 10 minutes before starting canine retraction stage; T1: 30 days following the onset of canine retraction; T2: 60 days; T3: 90 days following canine retraction onset; TF: At completion of canine retraction (expected to occur within 3-5 months)
  Anchorage loss is assessed by measuring first-molar movement relative to the third palatal ruga. Linear distances between the maxillary first molar fossa and the medial end of the third palatal ruga, both projected onto the mid-palatal plane, are recorded at T0-TF. Monthly drift rates are calculated similarly to canine retraction, averaged per side, and then across the cohort.
Change in Canine Angulation | T0: 10 minutes before starting canine retraction stage; T1: 30 days following the onset of canine retraction; T2: 60 days; T3: 90 days following canine retraction onset; TF: At completion of canine retraction (expected to occur within 3-5 months)
  Canine angulation change is evaluated at T0 and TF via standardized lateral cephalograms. To enhance measurement accuracy, stainless-steel reference wires (0.021 × 0.025 mm; 12 mm apical extension) are affixed to each canine: circular-ended on the right, triangular-ended on the left. Radiographs are analyzed in ImageJ (NIH, USA). Angulation is defined as the angle between each wire and the Sella-Nasion plane.
Root Resorption of the Canine | T0: T0: 10 minutes before starting canine retraction stage; TF: At completion of canine retraction (expected to happen within 3 - 5 months)
  External apical root resorption (EARR) is assessed by comparing maxillary canine root lengths on panoramic radiographs taken at T0 and TF. Baseline root length is recorded at T0; at TF, the reduction in length is measured, and the percentage of resorption is calculated. All measurements are performed in ImageJ (National Institutes of Health, Bethesda, Maryland, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad N. Kheshfeh, DDS, MSc, Principal Investigator — Department of Orthodontics, University of Damascus; Mohammad Younis Hajeer, DDS, MSc, PhD, Study Chair — Department of Orthodontics, University of Damascus; Ahamd S. Burhan, DDS, MSc, PhD, Study Director — Department of Orthodontics, Unviersity of Damascus
Locations (1):
- Orthodontics Department, Faculty of Dentistry, Damascus, Rif-dimashq Governorate, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mavreas D, Athanasiou AE. Factors affecting the duration of orthodontic treatment: a systematic review. Eur J Orthod. 2008 Aug;30(4):386-95. doi: 10.1093/ejo/cjn018. PMID 18678758
- [Background] Al-Ibrahim HM, Hajeer MY, Burhan AS, Sultan K, Ajaj MA, Mahaini L. The Efficacy of Accelerating Orthodontic Tooth Movement by Combining Self-Ligating Brackets With One or More Acceleration Methods: A Systematic Review. Cureus. 2022 Dec 23;14(12):e32879. doi: 10.7759/cureus.32879. eCollection 2022 Dec. PMID 36578856
- [Background] Kusy RP, Whitley JQ. Influence of archwire and bracket dimensions on sliding mechanics: derivations and determinations of the critical contact angles for binding. Eur J Orthod. 1999 Apr;21(2):199-208. doi: 10.1093/ejo/21.2.199. PMID 10327744
- [Background] Southard TE, Marshall SD, Grosland NM. Friction does not increase anchorage loading. Am J Orthod Dentofacial Orthop. 2007 Mar;131(3):412-4. doi: 10.1016/j.ajodo.2006.09.037. PMID 17346599
- [Background] Tidy DC. Frictional forces in fixed appliances. Am J Orthod Dentofacial Orthop. 1989 Sep;96(3):249-54. doi: 10.1016/0889-5406(89)90462-9. PMID 2773871